CLINICAL TRIAL: NCT00599339
Title: A Naturalistic, Multisite, Observational Study of Rotigotine Transdermal Patch and Other Currently Prescribed Therapies in Patients With Idiopathic Parkinson's Disease
Brief Title: Transdermal Rotigotine User Surveillance Study
Acronym: TRUST
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP0854
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2015-07

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Rotigotine; Neupro
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Neupro: Neupro at study onset
- Dopamine Agonist: Other Dopamine-Agonist at study onset
- L-Dopa: L-Dopa
- Neupro + L-Dopa: Neupro in combination with L-Dopa at study onset
- Dopamine Agonist + L-Dopa: Other Dopamine Agonist in combination with L-Dopa at study onset

SUMMARY:
This study will be conducted in an observational multiple-cohort design aimed at acquiring clinical, treatment, health status, and economic data. Patients with Parkinson's disease (PD) will be enrolled.

DETAILED DESCRIPTION:
All patients attending the physician and fulfilling the eligibility criteria are included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic early-stage Parkinson's Disease requiring dopaminergic monotherapy (rotigotine, other dopamine agonists or levodopa) at study onset
* Patients with advanced-stage Parkinson's Disease requiring dopaminergic therapy with levodopa in combination with rotigotine or other dopamine agonists at study onset

Exclusion Criteria:

* Patients who are unable to comply with study requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care
Sampling Method: Probability Sample
Enrollment: 2195 (Actual)
Dates: Start 2006-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (211):
- Czechia (14):
  - 813, Chomutov
  - 808, Hradec Králové
  - 822, Hradec Králové
  - 811, Litomyšl
  - 803, Ostrava-Poruba
  - 809, Pardubice
  - 817, Písek
  - 814, Plzen-Lochotin
  - 804, Prague
  - 805, Prague
  - 825, Prague
  - 829, Prague
  - 832, Rakovník
  - 819, Zlín
- Denmark (3):
  - 752, Aalborg
  - 751, Aarhus
  - 750, Sønderborg
- Germany (94):
  - 242, Aalen
  - 143, Achim
  - 240, Alzenau in Unterfranken
  - 145, Annaberg-Buchholz
  - 245, Aschaffenburg
  - 185, Augsburg
  - 130, Bad Neustadt an der Saale
  - 131, Bamberg
  - 103, Berg
  - 102, Berlin
  - 110, Berlin
  - 113, Berlin
  - 119, Berlin
  - 142, Berlin
  - 150, Berlin
  - 157, Berlin
  - 163, Berlin
  - 166, Berlin
  - 195, Berlin
  - 198, Berlin
  - 206, Berlin
  - 207, Berlin
  - 224, Berlin
  - 243, Berlin
  - 108, Bielefeld
  - 127, Bielefield
  - 178, Blankenburg (Harz)
  - 149, Bochum
  - 151, Bochum
  - 216, Bochum
  - 203, Böblingen
  - 220, Brandenburg
  - 236, Butzbach
  - 237, Butzbach
  - 124, Cologne
  - 153, Cologne
  - 179, Cologne
  - 133, Dresden
  - 199, Dresden
  - 232, Dresden
  - 219, Duisburg
  - 112, Düsseldorf
  - 141, Düsseldorf
  - 152, Eisleben Lutherstadt
  - 129, Emmendingen
  - 162, Erbach im Odenwald
  - 202, Flensburg
  - 156, Friedberg (Hessen)
  - 247, Gera
  - 223, Greifswald
  - 249, Hagen
  - 167, Halle
  - 121, Hamburg
  - 140, Hamburg
  - 176, Hamburg
  - 217, Hamburg
  - 241, Heidenheim
  - 138, Hemmoor
  - 173, Herborn
  - 214, Jena
  - 248, Jena
  - 181, Jülich
  - 105, Karlstadt am Main
  - 106, Karlstadt am Main
  - 244, Kassel
  - 175, Leutkirch
  - 230, Magdeburg
  - 235, Mannheim
  - 148, München
  - 189, München
  - 191, München
  - 169, Naumburg
  - 182, Neuburg am Inn
  - 118, Oberhausen
  - 164, Oberursel (Taunus)
  - 171, Oldenburg
  - 196, Oranienburg
  - 114, Rheda-Wiedenbrück
  - 188, Rottenburg Am Neckar
  - 187, Schriesheim
  - 107, Schwerin
  - 134, Singen
  - 229, Stadtroda
  - 180, Starnberg
  - 146, Stuttgart
  - 186, Stuttgart
  - 211, Stuttgart
  - 226, Tübingen
  - 139, Ulm
  - 172, Unterhaching
  - 239, Westerstede
  - 233, Wiesbaden
  - 122, Wolfach
  - 194, Zwickau
- Greece (10):
  - 607, Alexandroupoli
  - 600, Athens
  - 602, Athens
  - 605, Athens
  - 610, Athens
  - 608, Chaïdári
  - 611, Marousi
  - 601, Melíssia
  - 604, Thessaloniki
  - 606, Thessaloniki
- Italy (16):
  - 664, Acquaviva delle Fonti
  - 654, Ancona
  - 665, Bari
  - 655, Cagliari
  - 666, Casarano
  - 662, Cassino
  - 653, Ferrara
  - 661, Imperia
  - 650, Lido di Camaiore
  - 663, Lodi
  - 658, Messina
  - 660, Napoli
  - 667, Pisa
  - 657, Roma
  - 656, San Giovannni Rotondo
  - 669, Torino
- Mexico (9):
  - 704, Aguascalientes
  - 707, Guadalajara
  - 701, Mexico City
  - 702, Mexico City
  - 703, Mérida
  - 706, Monterrey
  - 710, Morelia Michoacan
  - 708, San Luis Potosí City
  - 705, Zapopan
- Romania (32):
  - 425, Arad
  - 406, Bacau
  - 407, Bacau
  - 417, Bistriţa
  - 412, Bucharest
  - 418, Bucharest
  - 423, Bucharest
  - 424, Bucharest
  - 434, Bucharest
  - 436, Bucharest
  - 427, Constanța
  - 411, Craiova
  - 433, Craiova
  - 404, Drobeta-Turnu Severin
  - 437, Foscani, Jud. Vrancea
  - 405, Galati
  - 420, Galati
  - 403, Lasi
  - 409, Lasi
  - 415, Medgidia
  - 402, Orăştie
  - 401, Piteşti
  - 428, Piteşti
  - 435, Râmnicu Vâlcea
  - 422, Resista
  - 408, Satu Mare
  - 429, Sfântu Gheorghe
  - 413, Sibiu
  - 416, Târgovişte
  - 432, Târgu Mureş
  - 414, Timișoara
  - 421, Timișoara
- Slovakia (16):
  - 521, Banská Bystrica
  - 500, Bratislava
  - 502, Bratislava
  - 507, Bratislava
  - 514, Bratislava
  - 501, Dolný Kubín
  - 505, Dubnica nad Váhom
  - 522, Krompachy
  - 520, Lučenec
  - 508, Skalica
  - 503, Spišská Nová Ves
  - 509, Stará Ľubovňa
  - 510, Trenčín
  - 519, Vranov nad Topľou
  - 518, Zvolen
  - 516, Žilina
- Spain (12):
  - 308, Alzira (Valencia)
  - 320, Badalona
  - 301, Barcelona
  - 303, Barcelona
  - 305, Barcelona
  - 318, Barcelona
  - 315, Burgos
  - 313, Ciudad Real
  - 306, Madrid
  - 307, Madrid
  - 314, Palma de Mallorca
  - 312, Valencia
- Switzerland (5):
  - 355, Biel
  - 354, Sankt Gallen
  - 353, Sargans
  - 351, Tschugg
  - 350, Zurich

REFERENCES:
- [Result] Muller T, Tolosa E, Badea L, Asgharnejad M, Grieger F, Markowitz M, Nondonfaz X, Bauer L, Timmermann L. An observational study of rotigotine transdermal patch and other currently prescribed therapies in patients with Parkinson's disease. J Neural Transm (Vienna). 2018 Jun;125(6):953-963. doi: 10.1007/s00702-018-1860-x. Epub 2018 Feb 26. PMID 29484495
- See also: Product Information — https://www.neupro.com/neupro-prescribing-information.pdf?v=1489766618
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll subjects in June 2006. Overall, 2195 patients were enrolled in this study (Enrolled Set [ES]), of which 2179 were treated with rotigotine or another Parkinson's disease treatment according to the study protocol at least once (Safety Set [SS]).
Pre-assignment Details: There were 36 patients without valid data consent. Therefore only Safety data were analyzed for these 36 patients.
  Patients without valid data consent or an unknown study termination status were neither considered as completer nor as non-completer in the Clinical Study Report. These patients are considered as non-completers in the summary below.
Groups:
- Overall: For this study, 5 groups of patients with different Parkinson's disease treatments were to be considered. Initial treatments were to include dopaminergic monotherapy with rotigotine, other dopamine agonists (eg, pramipexole, cabergoline, ropinirole), or L-dopa, treatment with L-dopa combined with rotigotine or other dopamine agonists. Treatment was to be performed according to standard medical practice. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
Period: Overall Study
Arm/Group | Overall
Started | 2195
Safety Set | 2179
Completed | 1531
Not Completed | 664
Not completed — Adverse Event | 79
Not completed — Withdrawal by Subject | 137
Not completed — Other Reason | 179
Not completed — Lost to Follow-up | 221
Not completed — No valid data consent | 36
Not completed — Study Termination Status Unknown | 12

BASELINE CHARACTERISTICS:
Population: Baseline Characterisitcs refer to the Enrolled Set [ES]. 2195 patients were enrolled in this study, of which 36 patients had no valid data consent. Data from these patients were not used for analysis.
Arm/Group | Overall
Number analyzed (Participants) | 2159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 724
  >=65 years | 1435
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 956
  Male | 1203

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part III at Visit 7 (Month 33)
Description: The Unified Parkinson's disease rating scale (UPDRS) Part III (Motor Examination) contains 31 questions. Each question ranges from 0 (best possible outcome) to 4 (worst outcome). The total score ranges from 0 (best possible outcome) to 124 (worst outcome).
Time Frame: From Baseline to Visit 7 (Month 33)
Population: All enrolled and treated patients, having at least one valid on-treatment measurement in any efficacy variable are included in the Full Analysis Set (FAS).
  Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Neupro Monotherapy (>= 3 Months): This group shows all subjects which were treated with Neupro for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with Neupro at Baseline.
- Neupro Monotherapy (< 3 Months): This group shows all subjects which were treated with Neupro for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with Neupro at Baseline.
- Other Dopamine Agonist (>= 3 Months): This group shows all subjects which were treated with other dopamine agonist for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with other dopamine agonist at Baseline.
- Other Dopamine Agonist (< 3 Months): This group shows all subjects which were treated with other dopamine agonist for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with other dopamine agonist at Baseline.
- L-Dopa Monotherapy (>= 3 Months): This group shows all subjects which were treated with L-Dopa for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with L-Dopa at Baseline.
- L-Dopa Monotherapy (< 3 Months): This group shows all subjects which were treated with L-Dopa for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with L-Dopa at Baseline.
- Multiple Dopamine Agonists (>= 3 Months): This group shows all subjects which were treated with multiple dopamine agonists for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with multiple dopamine agonists at Baseline.
- Multiple Dopamine Agonists (< 3 Months): This group shows all subjects which were treated with multiple dopamine agonists for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with multiple dopamine agonists at Baseline.
- Neupro + L-Dopa (>= 3 Months): This group shows all subjects which were treated with Neupro and L-Dopa for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with Neupro and L-Dopa at Baseline.
- Neupro + L-Dopa (< 3 Months): This group shows all subjects which were treated with Neupro and L-Dopa for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with Neupro and L-Dopa at Baseline.
- Other Dopamine Agonist + L-Dopa (>= 3 Months): This group shows all subjects which were treated with other dopamine agonist and L-Dopa for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with other dopamine agonist and L-Dopa at Baseline.
- Other Dopamine Agonist + L-Dopa (< 3 Months): This group shows all subjects which were treated with other dopamine agonist and L-Dopa for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with other dopamine agonist and L-Dopa at Baseline.
- Multiple Dopamine Agonists + L-Dopa (>= 3 Months): This group shows all subjects which were treated with multiple dopamine agonists and L-Dopa for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with multiple dopamine agonists and L-Dopa at Baseline.
- Multiple Dopamine Agonists + L-Dopa (< 3 Months): This group shows all subjects which were treated with multiple dopamine agonists and L-Dopa for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily treated with multiple dopamine agonists and L-Dopa at Baseline.
- Not Treated (>= 3 Months): This group shows all subjects which were not treated for 3 months or more at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily not treated at Baseline.
- Not Treated (< 3 Months): This group shows all subjects which were not treated for less than 3 months at Visit 7. Patients were to be given a treatment for Parkinson's disease deemed appropriate by the physician, and the treatment could be modified by the physician at any time during the study.
  Thus, subjects presented in this group weren't necessarily not treated at Baseline.
Arm/Group | Neupro Monotherapy (>= 3 Months) | Neupro Monotherapy (< 3 Months) | Other Dopamine Agonist (>= 3 Months) | Other Dopamine Agonist (< 3 Months) | L-Dopa Monotherapy (>= 3 Months) | L-Dopa Monotherapy (< 3 Months) | Multiple Dopamine Agonists (>= 3 Months) | Multiple Dopamine Agonists (< 3 Months) | Neupro + L-Dopa (>= 3 Months) | Neupro + L-Dopa (< 3 Months) | Other Dopamine Agonist + L-Dopa (>= 3 Months) | Other Dopamine Agonist + L-Dopa (< 3 Months) | Multiple Dopamine Agonists + L-Dopa (>= 3 Months) | Multiple Dopamine Agonists + L-Dopa (< 3 Months) | Not Treated (>= 3 Months) | Not Treated (< 3 Months)
Number analyzed (Participants) | 203 | 11 | 145 | 10 | 233 | 23 | 13 | 2 | 400 | 6 | 377 | 11 | 35 | 2 | 13 | 36
units on a scale | -2.5 (14.7) | -2.5 (10.3) | -2.2 (11.1) | -5.6 (16.9) | 0.2 (13.2) | 0.0 (12.2) | -1.2 (13.8) | 3.5 (6.4) | -1.2 (14.2) | -1.5 (17.5) | -2.5 (13.9) | 8.6 (13.5) | 1.5 (14.7) | 20.0 (29.7) | -3.2 (10.8) | 4.1 (15.0)

2. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Question 32 of Part IV at Visit 7 (Month 33)
Description: The Unified Parkinson's disease rating scale (UPDRS) question 32 of part IV asks. "What Proportion of the waking day are dyskinesias present?" Answers range from 0 (None) to 4 (76-100 % of the day).
Time Frame: From Baseline to Visit 7 (Month 33)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro Monotherapy (>= 3 Months) | Neupro Monotherapy (< 3 Months) | Other Dopamine Agonist (>= 3 Months) | Other Dopamine Agonist (< 3 Months) | L-Dopa Monotherapy (>= 3 Months) | L-Dopa Monotherapy (< 3 Months) | Multiple Dopamine Agonists (>= 3 Months) | Multiple Dopamine Agonists (< 3 Months) | Neupro + L-Dopa (>= 3 Months) | Neupro + L-Dopa (< 3 Months) | Other Dopamine Agonist + L-Dopa (>= 3 Months) | Other Dopamine Agonist + L-Dopa (< 3 Months) | Multiple Dopamine Agonists + L-Dopa (>= 3 Months) | Multiple Dopamine Agonists + L-Dopa (< 3 Months) | Not Treated (>= 3 Months) | Not Treated (< 3 Months)
Number analyzed (Participants) | 204 | 11 | 145 | 10 | 233 | 23 | 13 | 2 | 400 | 6 | 377 | 11 | 35 | 2 | 13 | 37
units on a scale | -0.1 (0.7) | -0.2 (0.6) | -0.1 (0.5) | 0.0 (0.8) | 0.1 (0.8) | -0.1 (0.5) | -0.1 (0.5) | 0.0 (0.0) | 0.1 (0.7) | 0.2 (1.0) | 0.2 (0.7) | 0.2 (0.6) | 0.2 (0.7) | 0.5 (0.7) | -0.2 (0.4) | 0.1 (0.8)

3. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Question 33 of Part IV at Visit 7 (Month 33)
Description: The Unified Parkinson's disease rating scale (UPDRS) Part IV question 33 asks for complications of therapy in the past week, through the question "How disabling are the dyskinesias ? " Answers range from 0 (Not disabling) to 4 (Completely disabling).
Time Frame: From Baseline to Visit 7 (Month 33)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro Monotherapy (>= 3 Months) | Neupro Monotherapy (< 3 Months) | Other Dopamine Agonist (>= 3 Months) | Other Dopamine Agonist (< 3 Months) | L-Dopa Monotherapy (>= 3 Months) | L-Dopa Monotherapy (< 3 Months) | Multiple Dopamine Agonists (>= 3 Months) | Multiple Dopamine Agonists (< 3 Months) | Neupro + L-Dopa (>= 3 Months) | Neupro + L-Dopa (< 3 Months) | Other Dopamine Agonist + L-Dopa (>= 3 Months) | Other Dopamine Agonist + L-Dopa (< 3 Months) | Multiple Dopamine Agonists + L-Dopa (>= 3 Months) | Multiple Dopamine Agonists + L-Dopa (< 3 Months) | Not Treated (>= 3 Months) | Not Treated (< 3 Months)
Number analyzed (Participants) | 204 | 11 | 145 | 10 | 233 | 23 | 13 | 2 | 400 | 6 | 377 | 11 | 35 | 2 | 13 | 37
units on a scale | -0.1 (0.7) | -0.2 (0.4) | -0.1 (0.4) | -0.1 (0.7) | 0.0 (0.8) | -0.0 (0.7) | -0.1 (0.6) | 0.0 (0.0) | 0.0 (0.7) | 0.0 (0.6) | 0.1 (0.7) | -0.1 (0.7) | 0.2 (0.8) | 0.0 (0.0) | -0.1 (0.3) | 0.2 (0.6)

4. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Question 39 of Part IV at Visit 7 (Month 33)
Description: The Unified Parkinson's disease rating scale (UPDRS) Part IV question 39 asks "What proportion of the waking day is the patient "off", on average?" Answers range from 0 (None) to 4 (76-100 % of the day).
Time Frame: 33 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro Monotherapy (>= 3 Months) | Neupro Monotherapy (< 3 Months) | Other Dopamine Agonist (>= 3 Months) | Other Dopamine Agonist (< 3 Months) | L-Dopa Monotherapy (>= 3 Months) | L-Dopa Monotherapy (< 3 Months) | Multiple Dopamine Agonists (>= 3 Months) | Multiple Dopamine Agonists (< 3 Months) | Neupro + L-Dopa (>= 3 Months) | Neupro + L-Dopa (< 3 Months) | Other Dopamine Agonist + L-Dopa (>= 3 Months) | Other Dopamine Agonist + L-Dopa (< 3 Months) | Multiple Dopamine Agonists + L-Dopa (>= 3 Months) | Multiple Dopamine Agonists + L-Dopa (< 3 Months) | Not Treated (>= 3 Months) | Not Treated (< 3 Months)
Number analyzed (Participants) | 204 | 11 | 145 | 10 | 233 | 23 | 13 | 2 | 400 | 6 | 377 | 11 | 35 | 2 | 13 | 37
units on a scale | -0.2 (0.9) | 0.5 (0.9) | -0.1 (0.8) | 0.1 (0.9) | 0.1 (0.9) | 0.1 (1.1) | -0.4 (0.9) | 0.0 (0.0) | 0.0 (0.8) | 0.0 (0.0) | 0.2 (0.9) | 0.2 (0.9) | -0.0 (1.0) | 1.5 (2.1) | 0.0 (0.4) | 0.3 (0.9)

5. Secondary Outcome: Change From Baseline in Nocturnal Dystonia Cramp Score (NADCS) at Visit 7 (Month 33)
Description: The NADCS assesses sleep-related motor complaints including nocturnal akinesia, dystonia and painful cramps by an ordinal severity scale.
  The NADCS total score ranges from 0 (normal) to 4 (maximum severity). NADCS value was missing for one subject at Visit 7.
Time Frame: 33 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro Monotherapy (>= 3 Months) | Neupro Monotherapy (< 3 Months) | Other Dopamine Agonist (>= 3 Months) | Other Dopamine Agonist (< 3 Months) | L-Dopa Monotherapy (>= 3 Months) | L-Dopa Monotherapy (< 3 Months) | Multiple Dopamine Agonists (>= 3 Months) | Multiple Dopamine Agonists (< 3 Months) | Neupro + L-Dopa (>= 3 Months) | Neupro + L-Dopa (< 3 Months) | Other Dopamine Agonist + L-Dopa (>= 3 Months) | Other Dopamine Agonist + L-Dopa (< 3 Months) | Multiple Dopamine Agonists + L-Dopa (>= 3 Months) | Multiple Dopamine Agonists + L-Dopa (< 3 Months) | Not Treated (>= 3 Months) | Not Treated (< 3 Months)
Number analyzed (Participants) | 204 | 11 | 145 | 10 | 232 | 23 | 13 | 2 | 400 | 6 | 376 | 11 | 34 | 2 | 13 | 37
units on a scale | -0.27 (1.79) | 1.36 (3.51) | -0.15 (1.48) | 0.05 (2.53) | -0.09 (1.84) | -0.26 (2.30) | -0.73 (1.49) | 0.75 (1.06) | -0.03 (2.06) | -0.42 (2.01) | -0.03 (2.07) | 1.05 (1.39) | -0.01 (1.90) | 3.25 (4.60) | -0.38 (1.10) | 0.22 (2.19)

6. Secondary Outcome: Hoehn & Yahr Stage at Visit 7 (Month 33)
Description: The Hoehn and Yahr staging of Parkinson's disease in the "on" stage, if applicable, had to be completed by the physician.
  Possible staging:
  * 0 No signs of disease
  * 1 Unilateral disease
  * 2 Bilateral disease without impairment of balance
  * 3 Mild to moderate bilateral disease, some postural instability, physically dependent
  * 4 Severe disability, still able to walk or stand unassisted
  * 5 Wheelchair bound or bedridden unless aided
Time Frame: 33 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Neupro Monotherapy (>= 3 Months) | Neupro Monotherapy (< 3 Months) | Other Dopamine Agonist (>= 3 Months) | Other Dopamine Agonist (< 3 Months) | L-Dopa Monotherapy (>= 3 Months) | L-Dopa Monotherapy (< 3 Months) | Multiple Dopamine Agonists (>= 3 Months) | Multiple Dopamine Agonists (< 3 Months) | Neupro + L-Dopa (>= 3 Months) | Neupro + L-Dopa (< 3 Months) | Other Dopamine Agonist + L-Dopa (>= 3 Months) | Other Dopamine Agonist + L-Dopa (< 3 Months) | Multiple Dopamine Agonists + L-Dopa (>= 3 Months) | Multiple Dopamine Agonists + L-Dopa (< 3 Months) | Not Treated (>= 3 Months) | Not Treated (< 3 Months)
Number analyzed (Participants) | 207 | 11 | 146 | 11 | 234 | 23 | 13 | 2 | 401 | 6 | 378 | 11 | 36 | 2 | 13 | 37
participants
  0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  1 | 55 | 1 | 48 | 0 | 29 | 1 | 0 | 1 | 29 | 2 | 37 | 0 | 2 | 0 | 4 | 3
  2 | 112 | 4 | 76 | 6 | 118 | 12 | 7 | 1 | 186 | 2 | 192 | 2 | 15 | 1 | 7 | 19
  3 | 28 | 4 | 19 | 4 | 70 | 8 | 5 | 0 | 131 | 2 | 119 | 4 | 13 | 0 | 1 | 11
  4 | 8 | 2 | 2 | 0 | 14 | 2 | 1 | 0 | 46 | 0 | 24 | 4 | 3 | 1 | 1 | 3
  5 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 6 | 0 | 4 | 1 | 2 | 0 | 0 | 1
  No Data/Missing | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0

7. Secondary Outcome: Reported Adverse Events of Cardiac Valve Fibrosis During the Study (up to 33 Months)
Description: The analysis was performed for the non-disjunctive classification into patients at risk to develop an Adverse Event associated with Rotigotine and patients at risk to develop an Adverse Event not associated with Rotigotine.
Time Frame: 33 months
Population: For analysis of Safety the patients in the Safety Set were sub-grouped into patients at risk developing an Adverse Event (AE) associated with rotigotine and patients at risk developing an AE not associated with rotigotine. This sub-grouping is non-disjunctive in nature, i.e. one patient might fall into both subgroups.
Measure: Number; unit: Adverse Events
Groups:
- Associated With Rotigotine: A patient was analyzed related to Adverse Events (AEs) associated with Rotigotine only if during the study he was at risk to develop an AE associated with Rotigotine.
  An Adverse Event was considered to be associated with Rotigotine if Rotigotine was administered at least once within 30 days prior to the onset of the adverse event. "Associated Event" does not necessarily mean related to treatment with Rotigotine.
- Not Associated With Rotigotine: A patient was analyzed related to Adverse Events (AEs) not associated with Rotigotine only if during the study he was at risk to develop an AE not associated with Rotigotine.
  An adverse event was considered not to be associated with Rotigotine, if no Rotigotine was administered in the 30 days period prior to the onset of the AE.
Arm/Group | Associated With Rotigotine | Not Associated With Rotigotine
Number analyzed (Participants) | 1390 | 1328
Adverse Events
  Cardiac valve disease | 1 | 1
  Cardiac valve sclerosis | 0 | 2
  Aortic valve sclerosis | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected during the course of the study from Baseline (Visit 1) up to Visit 7 (Month 33 ± 30 days).
Description: For analysis of Safety the patients in the Safety Set were sub-grouped into patients at risk developing an Adverse Event (AE) associated with rotigotine and patients at risk developing an AE not associated with rotigotine. This sub-grouping is non-disjunctive in nature, i.e. one patient might fall into both subgroups.
Arm/Group | Associated With Rotigotine | Not Associated With Rotigotine
Serious Adverse Events (participants affected / at risk) | 261/1390 | 269/1328
Other Adverse Events (participants affected / at risk) | 237/1390 | 245/1328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Associated With Rotigotine (N=1390) | Not Associated With Rotigotine (N=1328)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 7 (7) | 7 (7)
Angina pectoris (Cardiac disorders) | 3 (3) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (5) | 9 (9)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory distress (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 4 (4)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery restenosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block third degree (Cardiac disorders) | 3 (3) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 3 (3)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve sclerosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Acromegaly (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 7 (7) | 5 (5)
Sudden death (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 3 (3) | 2 (2)
Orthostatic intolerance (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Application site rash (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 8 (8)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngotracheo bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Norwalk virus (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Mycotoxicosis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 8 (9)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pharyngeal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vertebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Investigation (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (11)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (10)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (6)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 39 (47) | 32 (38)
Parkinsonism (Nervous system disorders) | 1 (1) | 2 (3)
Ischaemic stroke (Nervous system disorders) | 8 (8) | 7 (7)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 4 (6)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 9 (9) | 4 (5)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 4 (4) | 5 (5)
Progressive supranuclear palsy (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 4 (4)
Cerebral hypoperfusion (Nervous system disorders) | 0 (0) | 1 (1)
Hypokinesia (Nervous system disorders) | 2 (2) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 2 (2)
Fine motor delay (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Pseudoradicular syndrome (Nervous system disorders) | 2 (2) | 1 (1)
Spinal cord haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 2 (2)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Phrenic nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonic epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (2)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Drop attacks (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 8 (8)
Hallucination (Psychiatric disorders) | 2 (2) | 2 (2)
Hallucination, visual (Psychiatric disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep attacks (Psychiatric disorders) | 2 (2) | 0 (0)
Somatoform disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cyclothymic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Binge eating (Psychiatric disorders) | 0 (0) | 1 (1)
Impulse-control disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hypersexuality (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Therapy regimen changed (Surgical and medical procedures) | 3 (3) | 1 (1)
Device therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug therapy changed (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep brain stimulation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2)
Varicose ulceration (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (2) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Associated With Rotigotine (N=1390) | Not Associated With Rotigotine (N=1328)
Nausea (Gastrointestinal disorders) | 105 (120) | 85 (101)
Fatigue (General disorders) | 67 (76) | 77 (82)
Fall (Injury, poisoning and procedural complications) | 49 (60) | 67 (79)
Depression (Psychiatric disorders) | 54 (55) | 72 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days